CLINICAL TRIAL: NCT02356718
Title: Cognitive Training in Inpatient Treatment for Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Christian Hendershot, Assistant Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0422014
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Computerized cognitive training activities
  Interventions: Behavioral: Cognitive training activities; Behavioral: Inpatient psychosocial therapy
- Control (Active Comparator): Non-adaptive computerized cognitive training activities
  Interventions: Behavioral: Cognitive training activities; Behavioral: Inpatient psychosocial therapy

INTERVENTIONS:
Behavioral: Cognitive training activities — Training activities consist of computer tasks designed to improve memory and cognition. The intervention consists of 45-minute training sessions delivered regularly during inpatient treatment.
Behavioral: Inpatient psychosocial therapy — Group psychosocial therapy delivered in an inpatient setting.

SUMMARY:
This study examines whether computer tasks can improve memory and other cognitive functions among patients receiving inpatient treatment for substance use disorders.

DETAILED DESCRIPTION:
Participants will complete cognitive training sessions on a regular basis during inpatient treatment. Alternate versions of the computer tasks will be compared in a randomized design. Primary and secondary outcomes will consist of changes in cognitive performance before and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be patients registered for inpatient treatment at the Centre for Addiction and Mental Health
* Age 18-60
* Fluency in English
* Able to attend scheduled training sessions
* Comfortable using a computer and mouse

Exclusion Criteria:

* Severe cognitive impairment
* Current or past psychosis or diagnosis of schizophrenia
* Photosensitive epilepsy or history of seizures triggered by light
* Legal mandate to attend treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Auditory memory capacity - WAIS Digit Span score | Baseline, 3 weeks
  WAIS Digit Span score

SECONDARY OUTCOMES:
Auditory memory capacity - WAIS Letter-number sequencing score | Baseline to 3 weeks
  WAIS Letter-number sequencing score
Visual memory capacity - WMS Spatial span score | Baseline to 3 weeks
  WMS Spatial span score
Visual memory capacity - WMS Symbol span score | Baseline to 3 weeks
  WMS Symbol span score
Training progress score - Cognitive progress indicator score | Baseline to 4 weeks
  Cognitive progress indicator score

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hendershot, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hendershot CS, Wardell JD, Vandervoort J, McPhee MD, Keough MT, Quilty LC. Randomized trial of working memory training as an adjunct to inpatient substance use disorder treatment. Psychol Addict Behav. 2018 Dec;32(8):861-872. doi: 10.1037/adb0000415. Epub 2018 Nov 26. PMID 30475014
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research